CLINICAL TRIAL: NCT05107713
Title: Positioning of EDI Catheter In Premature Infants
Acronym: PIPI
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 21-078
Record Dates: First submitted 2021-10-25; First posted 2021-11-04 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Evaluation of Preterm NAVA Catheter Placement
Keywords: Neurally Adjusted Ventilatory Assist, NAVA catheter, Edi catheter, electrical activity of the diaphragm, feeding tube placement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Nasogastric (NG) and orogastric (OG) feeding tubes have a high incidence of malpositioning, occurring in up to 59% of preterm infants (Lopes 2019). Ideally, the tip of the feeding tube (including the orifices) should be located within the body of the stomach.

Malpositioning of the feeding tube can be classified as (i) being "too far out" where the tip of the catheter is located in the esophagus above the gastro-esophageal junction, potentially resulting in reflux, aspiration, apnea or (ii) being inserted "too far in" where the tip is located in the pylorus or the duodenum, leading to malabsorption of nutrients, diarrhea, and poor weight gain. Feeding tubes can also be found "curled up" inside the stomach (Quandt 2009) as much as 35% of the time. As well, one cannot ignore the risk of perforation, where the incidence has been reported to be 1.1% in extremely low birth weight (ELBW) infants (<1000g) (n = 7/646) (Thanhaeuser M, 2019); of note: perforations occurred on the third day of life (range days 2-14) not during initial feeding tube placement.

In 2008, a modified feeding tube was introduced to the market (Maquet Critical Care AB), which contains sensors placed in its wall, 13 mm above the feeding orifices, used for measuring the electrical activity of the diaphragm (Edi) during spontaneous breathing. The Edi signal is then used to neurally control mechanical ventilation, or for neural monitoring of the breathing pattern (Sinderby 1999; Beck 2016). The so-called "Edi catheter" comes with the manufacturer's recommended insertion measurements and verification window. In the Servo-I, the insertion distance is provided by a formula on the catheter packaging. In the Servo-U and Servo-n, the calculation for predicted insertion is provided by a tool in the ventilator. There is no available, published data upon which the manufacturer's recommendations were based. It is possible that obtaining appropriate positioning of the Edi catheter - based on a pattern of electrical signals from the sensors - could reduce the incidence of malposition.

This proposed study is observational, and non-interventional. The purpose is to verify the position of a neurally guided, clinically-placed, Edi catheter using radiography (Ellett 2011). We will also record physical measurements and weights of the babies in order to validate previously described methods of predicting insertion length. The x-rays will be taken with "near-simultaneous" screenshots of the Edi catheter positioning window.

DETAILED DESCRIPTION:
Nasogastric (NG) and orogastric (OG) feeding tubes have a high incidence of malpositioning, occurring in up to 59% of preterm infants (Lopes 2019). Ideally, the tip of the feeding tube (including the orifices) should be located within the body of the stomach.

Malpositioning of the feeding tube can be classified as (i) being "too far out" where the tip of the catheter is located in the esophagus above the gastro-esophageal junction, potentially resulting in reflux, aspiration, apnea or (ii) being inserted "too far in" where the tip is located in the pylorus or the duodenum, leading to malabsorption of nutrients, diarrhea, and poor weight gain. Feeding tubes can also be found "curled up" inside the stomach (Quandt 2009) as much as 35% of the time. As well, one cannot ignore the risk of perforation, where the incidence has been reported to be 1.1% in extremely low birth weight (ELBW) infants (<1000g) (n = 7/646) (Thanhaeuser M, 2019); of note: perforations occurred on the third day of life (range days 2-14) not during initial feeding tube placement.

In 2008, a modified feeding tube was introduced to the market (Maquet Critical Care AB), which contains sensors placed in its wall, 13 mm above the feeding orifices, used for measuring the electrical activity of the diaphragm (Edi) during spontaneous breathing. The Edi signal is then used to neurally control mechanical ventilation, or for neural monitoring of the breathing pattern (Sinderby 1999; Beck 2016). The so-called "Edi catheter" comes with the manufacturer's recommended insertion measurements and verification window. In the Servo-I, the insertion distance is provided by a formula on the catheter packaging. In the Servo-U and Servo-n, the calculation for predicted insertion is provided by a tool in the ventilator. There is no available, published data upon which the manufacturer's recommendations were based. It is possible that obtaining appropriate positioning of the Edi catheter - based on a pattern of electrical signals from the sensors - could reduce the incidence of malposition.

This proposed study is observational, and non-interventional. The purpose is to verify the position of a neurally guided, clinically-placed, Edi catheter using radiography (Ellett 2011). The investigators will also record physical measurements and weights of the babies in order to validate previously described methods of predicting insertion length. The x-rays will be taken with "near-simultaneous" screenshots of the Edi catheter positioning window.

The investigators plan on studying a convenience sample of 65 premature babies of varying weights, from 9 sites.

Objective of the study:

To determine if optimal positioning of the Edi catheter results in feeding holes in the stomach in neonates. The aim is to capture a screenshot of the Edi catheter positioning along with one radiograph.

Study design:

This is a multi-centre, observational study.

Procedures:

1. Once the subject is enrolled, if not already inserted, the Edi catheter will be placed as guided by routine clinical practice and fixed in place.
2. Data collection form will be completed.
3. When the placement of the Edi catheter is deemed satisfactory (or may have already been in place), a screenshot or photograph of the catheter positioning window is taken. Clinicians should make an effort to capture a screenshot just prior to or immediately after the radiograph is done, taking effort to maintain the same patient positioning to prevent inadvertent migration of the Edi catheter.
4. Radiograph taken.
5. Send all info to J Beck: package would include de-identified data: Data collection form, screen shot, radiograph.
6. De-identified data will be initially sent to a secure server at Neurovent Research Inc, for then transfer to St-Michael's Hospital (lead site).

Analysis:

Radiographs will be analyzed after-the-fact, by Dr. Kay North, without having information on the catheter positioning window. The location of the tip of the catheter will be classified into one of four categories: 1. Tube tip in esophagus. 2 Tube tip in the region of the GEJ. 3. Tube tip in the stomach. 4. Tube tip in the pylorus. Any other comments would be noted (e.g. curled up catheter, catheter tip impinging on the lateral gastric wall), (Quandt 2009).

Screenshot of positioning window. Two independent analysts from St-Michael's Hospital will determine diaphragm position on the array. With the 6 mm IED catheter we have a resolution of 12 mm.

The measurements on the data collection form about NEX, NEMU and ARHB will be correlated to catheter insertion distance.

Other data will be used for anthropometric information

ELIGIBILITY:
Inclusion Criteria:All babies, irrespective of GA, whose current weight is 400-2000g, who are:

* about to be equipped OR already equipped with a 6F or 8F (49 or 50 cm) Edi feeding tube for clinical or research purposes.
* Babies who are prescribed clinically or for research purposes, to have a chest/abdominal radiograph. Babies may be breathing on NAVA, NIV-NAVA or neural monitoring during a conventional mode or HFO, or nCPAP/HFNC.
* Placement of a second feeding tube is permitted, as well as oral or nasal feeding tube insertion.

Our goal is to study a minimum of 65 babies. We will try to obtain data from the following (6) weight categories with a minimum of 10 babies in each category, except the smallest group where we anticipate positioning to be more challenging, based on anatomical modelling:

400-750g (n= 15 babies) 750-1000g (n = 10 babies) 1000-1250g (n = 10 babies) 1250-1500g (n = 10 babies) 1500-1750g (n = 10 babies) 1750-2000g (n = 10 babies). The investigators are aware that not all centres use Edi catheters in all the different weight groups.

-

Exclusion Criteria:

Patient exclusion criteria:

Previous gastric surgery, anatomical abnormalities. Further reasons for exclusion will be left to the clinicians at each site.

-

Ages: 1 Day to 1 Year | Sex: All
Age Groups: Child
Study Population: All babies, irrespective of GA, whose current weight is 400-2000g, who are:
  * about to be equipped OR already equipped with a 6F or 8F (49 or 50 cm) Edi feeding tube for clinical or research purposes.
  * Babies who are prescribed clinically or for research purposes, to have a chest/abdominal radiograph. Babies may be breathing on NAVA, NIV-NAVA or neural monitoring during a conventional mode or HFO, or nCPAP/HFNC.
  * Placement of a second feeding tube is permitted, as well as oral or nasal feeding tube insertion
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
position of NAVA catheter determined by xray | 1 year
  Radiographs of clinically placed catheters will be evaluated by an independent radiologist

CONTACTS AND LOCATIONS:
Locations (1):
- Unity Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Radiographs will be analyzed by an independent radiologist
Supporting Information: Study Protocol
Time Frame: 1 year
Access Criteria: de-identified radiographs